CLINICAL TRIAL: NCT02921815
Title: Revlimid 5 mg Capsules Special Use-results Surveillance of Transformation to Acute Myeloid Leukemia
Brief Title: A Study to Analyze the Occurrence of Transformation From Myelodysplastic Syndrome to Acute Myeloid Leukemia in Patients With Myelodysplastic Syndrome Who Received Revlimid® 5 mg Capsules and Who Are Continuing or no Longer Continuing Revlimid Treatment
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-Celgene-JP-PMS-001c
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute
Keywords: Leukemia; Acute Myeloid Leukemia; Revlimid
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with myeloid leukemia: All del(5q) Myelodysplastic syndrome (MDS) patients in the all-case surveillance in whom transformation to acute myeloid leukemia has not been documented at the end of the observation period of the all-case surveillance.

SUMMARY:
To analyze the occurrence of transformation from myelodysplastic syndrome (MDS) to acute myeloid leukemia (hereinafter referred to as transformation from MDS to AML) in patients with myelodysplastic syndrome with a deletion 5q cytogenetic abnormality (hereinafter referred to as del(5q)MDS) who received Revlimid® 5 mg Capsules (hereinafter referred to as Revlimid) and who are continuing or no longer continuing Revlimid treatment.

1. Planned registration period This period started on the date of initial marketing of Revlimid and will end on the day when the appropriateness of enrollment is assessed for all del(5qMDS) patients in the all-case surveillance.
2. Planned surveillance period This period started on the date of initial marketing of Revlimid and will end 3 years after the last enrolled patient begins receiving Revlimid.

ELIGIBILITY:
Inclusion Criteria:

* All del(5q)MDS patients in the all-case surveillance in whom transformation to acute myeloid leukemia (hereinafter referred to as AML) has not been documented at the end of the observation period of the all-case surveillance.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All del(5q) Myelodysplastic syndrome (MDS) patients in the all-case surveillance in whom transformation to acute myeloid leukemia (hereinafter referred to as Acute Myelogenous Leukemia (AML)) has not been documented at the end of the observation period of the all-case surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 3 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Shinko Hospital, Kobe, Hyōgo, Japan